CLINICAL TRIAL: NCT06144619
Title: Non-Invasive Biomarkers in Prostate Cancer Disease Management
Status: Suspended | Type: Observational
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22098
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Intermediate Risk Prostate Cancer; High Risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intermediate risk group (no-surgery): Participants diagnosed with pre-biopsy mpMRI.
  Interventions: Genetic: Genomic and Histological Evaluation
- High-risk group (surgery): Participants who had radical prostatectomy (RP) with (or with-out) mpMR imaging.
  Interventions: Genetic: Genomic and Histological Evaluation

INTERVENTIONS:
Genetic: Genomic and Histological Evaluation — Participants will obtain genomic and histological evaluation on their biopsied samples. (Follows SOC)

SUMMARY:
This study is an observational retrospective/ prospective study with diagnosed low/intermediate risk (no-surgery) & high risk (surgery) prostate cancer that are eligible and willing to undergo standard of care (SOC) assessment, annually along with biopsies, bio-fluid collection. Participants will obtain genomic and histological evaluation on their biopsied samples. Study follows SOC collection with additional body fluid collection (blood, urine). Biopsy/surgery will not require additional sample collection

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who had received primary diagnosis at Moffitt or outside the cancer center with available records (radiology, pathology, access to samples).
* No-Surgery (Intermediate risk) group: patients diagnosed with pre-biopsy mpMRI, blood plasma: the biopsy must consist of a pathological diagnosis with a Gleason pattern score.
* Surgery (High risk) group: patients who had radical prostatectomy (RP) with (or with-out) mpMR imaging, bio fluids available for research will be accrued for this group. We follow the NCCN recommendations for high-risk (Unfavorable intermediate risk or High-risk) groups inclusion and follow-up criteria (58, 89, 90).
* ≥ 4 ng/ml and ≤ 20 ng/ml and PSA ≤ 10 ng/ml (for late disease), within 3 months of study enrollment.
* Age 35 through 85 years.
* Zubrod/ECOG performance status <2;
* Ability to understand and willingness to sign a written informed consent document.
* Patients who agree to have a multiparametric MRI with targeted/template biopsy.
* Patients must agree to fill out the longitudinal psychosocial questionnaires assessing health related quality of life.
* Availability of Bio-samples (blood plasma, urine) for exosomal, proteomic, genomic and pathology (H&E slides, IHC slides).
* Quantity of bio-samples; Blood, Urine, tissue sections (including FFPE) for each region of interest.

Exclusion Criteria:

* Subject is not a candidate for multiparametric MRI with contrast. Some reasons may include (but are not limited to): renal insufficiency, foreign body or pacemakers.
* No prior pelvic radiotherapy
* No prior surgery to the prostate, other than transurethral procedures for benign prostatic hyperplasia (e.g., transurethral resection, green light laser treatment)
* No concurrent, active malignancy, other than non-metastatic skin cancer of any type, superficial bladder cancer, or early-stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma) or > Bilateral hip replacement.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients who had received primary diagnosis at Moffitt or outside the cancer center with available records (radiology, pathology, access to tissue samples).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | Up to 3 years
  Progression will be defined according to the National Comprehensive Cancer Network (NCCN) clinical guidelines.
  Intermediate risk group (no-surgery): Evaluation of targeted lesion indicates any one of the following: a) Gleason grade group of 2 or 3 (Gleason Score: 3+4 or 4+3), b) re-biopsy of lesion results in higher Gleason grade, initial GS 3+3 becomes a 3+4 or higher and c) secondary end point include clinical progression assessed by radiological progression (increased PIRADS score) and/or serum progression (PSA increase).
  High risk group (surgery): Participants who undergo prostatectomy as standard of care recommendation, following the NCCN guidelines. Participants in this group fall under these clinical characteristics: a) unfavorable intermediate-risk: biopsies with GS 4+3 or higher, b) high risk for prostate cancer progression: biopsies with GS 4+4 or greater or cT3 or greater disease, c) Progression following treatment, increase in PSA (

CONTACTS AND LOCATIONS:
Overall Officials: Yoganand Balagurunathan, PhD, Principal Investigator — Moffitt Cancer Center; Julio Pow-Sang, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No